CLINICAL TRIAL: NCT07159113
Title: The Relationship Between Sensory Profile and Ankle Muscle Shortness in Children With Autism
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor Dr., Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-10
Record Dates: First submitted 2025-05-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to investigate the relationship between sensory profile and ankle muscle shortness in children with autism.

This study will feature only one group consisting of children with autism

Childhood autism assessment scale will be completed with the families of the children included in the study. The tip-toe walking status of the children participating in the study will be observed and classified according to the tip-toe walking classification. The ankle muscle shortness of the children will be evaluated by Gastro-Soleus shortness measurements and sensory processing skills will be evaluated by Sensory profile.

Muscle shortness measurements and sensory profile results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with autism spectrum disorder in the Special Needs Report for Children (ÇÖZGER)
* GMFCS level I,II or III
* Between the ages of 4-10
* Volunteering to participate in the study

Exclusion Criteria:

* Having a rigid contracture in passive knee extension and ankle range of motion
* History of surgery or botox affecting ankle joint range of motion in the last 6 months

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study includes children with autism between the ages of 4-10
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Sensory Profile | One year
  This test is used to assess how children aged 3-10 years process information from their body and environment. It is a five-point Likert-type parent questionnaire and consists of 125 items. It is explained to the caregiver that he/she should check the box that best describes how often the child performs the behaviors given in the questionnaire and answer for all parameters; if he/she cannot answer because there is a behavior that he/she cannot observe at all or that he/she thinks does not fit the child, he/she should put an X on that question.
  The end of each section is scored according "always" 1, "frequently" 2, "occasionally" 3, "rarely" 4, "never" 5. The scores obtained from each parameter are calculated according to the Dunn Sensory Profile Score Explanation and the child is classified according to the categories of 'definite difference', 'probable difference', 'typical performance' from each section.

SECONDARY OUTCOMES:
Childhood Autism Rating Scale | One year
  It is a scale consisting of 15 items used to assess the severity of autism, with each item scored between 1 and 4. A score of 1 represents that the child's behavior for that item is normal for his/her age, while a score of 4 represents that it is extremely abnormal. The minimum score is 15 and the maximum score is 60. The results are evaluated as "no autism" between 15-29 points, "mild-moderate autism" between 30-36 points, and extreme autism between 37-60 points. Families of the children were asked to fill out the froms.
M.Gastrocnemius - M.Gastrosoleus Shortness Measurement | One year
  Passive foot dorsiflexion measurement with a manual goniometer was performed at 0 degrees knee flexion for Gastrocnemius muscle and 90 degrees knee flexion for Soleus muscle. Muscle shortness was expressed in degrees. Ankle neutral position was recorded as 0 degrees, dorsiflexion angles as positive and plantar flexion angles as negative.
Classification of Tiptoe Walking | One year
  Tiptoe walking was assessed and classified by observation during 10-meter walk-run. Level 1 indicates that there is tiptoe behavior during running, walking and standing; Level 2 indicates that there is tiptoe behavior during running and walking; Level 3 indicates that there is tiptoe behavior only during running; if no tiptoe walking is observed, it was indicated as "no tiptoe walking".

CONTACTS AND LOCATIONS:
Overall Officials: Seda Ayaz Taş, Phd, Principal Investigator — Abant Izzet Baysal University
Locations (3):
- Turkey (Türkiye) (3):
  - Bolu Abant İzzet Baysal University, Bolu, Bolu
  - Düzce Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Düzce, Düzce
  - Kdz. Ereğli Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Ereğli, Zonguldak Province

IPD SHARING:
Plan to Share IPD: No